CLINICAL TRIAL: NCT07325591
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Tazbentetol in Participants With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy and Safety of Tazbentetol in ALS Participants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPG302-ALS-003 (SPARK)
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: regenerative; synapse; Amyotrophic Lateral Sclerosis; placebo-controlled
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- tazbentetol 300 mg once daily (Experimental): synthetic small molecule
  Interventions: Drug: Tazbentetol 300 mg once daily; Drug: placebo
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- tazbentetol 300 mg twice daily (Experimental): synthetic small molecule
  Interventions: Drug: Tazbentetol 300 mg twice daily

INTERVENTIONS:
Drug: Tazbentetol 300 mg once daily — participants in double blind placebo controlled phase will be randomized to received study drug tazbentetol at 300 mg once daily and placebo tablets once daily. Participants in the open-label extension phase will receive the dose determined from DBPC.
  Other Names: SPG302
  Arms: tazbentetol 300 mg once daily
Drug: placebo — participants in double blind placebo controlled phase will be randomized to received placebo tablets twice daily.
  Arms: Placebo; tazbentetol 300 mg once daily
Drug: Tazbentetol 300 mg twice daily — participants in double blind placebo controlled phase will be randomized to received study drug tazbenetol at 300 mg twice daily. Participants in the open-label extension phase will receive the dose determined from DBPC.
  Other Names: SPG302
  Arms: tazbentetol 300 mg twice daily

SUMMARY:
The objectives of this study are to examine the effects of tazbentetol on clinical measures of ALS, patient reported outcomes (PROs), long-term safety and tolerability.

DETAILED DESCRIPTION:
This is a Phase 2b adaptive design randomized, double-blind, placebo-controlled (DBPC) study to evaluate the efficacy, safety and tolerability of tazbentetol administered orally in participants with ALS.

The study consists of 2 parts, as follows

Double-blind, placebo controlled (DBPC): Randomized, double-blind, placebo-controlled with 3 parallel treatments arms. Participants will be randomized in a 1:1:1 ratio to receive either tazbentetol 300 mg once daily (QD), or 300 mg twice daily (BID), or placebo for 36 weeks.

Open-label extension: Eligible participants who complete 36 weeks in the DBPC will be offered to enroll into the OLE, starting at the corresponding DBPC Week 36 visit, and receive tazbentetol for 36 weeks. The dose for this extension will be based on data from DBPC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* ALS TRICALS risk score
* Stable dose of standard of care treatment
* Contraception use by men or women consistent with local regulations
* Able and willing to provide written informed consent

Exclusion Criteria:

* Underlying physical or psychological condition prohibiting study completion
* Clinically significant cardiac disease
* Active or history of malignancy in the past 5 years
* Serious infection within 1 month of screening
* Acute illness within 30 days of Day 1
* History of suicidal behavior or suicidal ideation
* Active cigarette smokers and users of nicotine-containing products
* Neurodegenerative disease
* External respiratory support or supplemental oxygen requirement
* HIV, hepatitis B and hepatitis C positive
* Vaccines within 14 days
* Other investigational products within 30 days
* Blood donation within 30 days
* Plasma donation within 7 days
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale-revised (ALSFRS-R) total score | 36 weeks for DBPC
  Questionnaire administered by a clinician that measures participants' ability to function in certain daily activities. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Absolute change from baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale-revised (ALSFRS-R) total score | 36 weeks for OLE
  Questionnaire administered by a clinician that measures participants' ability to function in certain daily activities. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.

SECONDARY OUTCOMES:
Combined Assessment of Function and Survival (CAFS) scores | 36 weeks for DBPC
  This assessment ranks clinical outcome based on changes to ALSFRS-R score. A higher score indicates a better clinical outcome.
Combined Assessment of Function and Survival (CAFS) scores | 36 weeks for OLE
  This assessment ranks clinical outcome based on changes to ALSFRS-R score. A higher score indicates a better clinical outcome.
Change from baseline in Clinician Global Impression-Inhibitory (CGI-I) | 36 weeks for DBPC
  Change in clinician rated measures on scale of 1 to 7, higher value indicates more severe symptom presentation
Change from baseline in Clinician Global Impression-Inhibitory (CGI-I) | 36 weeks for OLE
  Change in clinician rated measures on scale of 1 to 7, higher value indicates more severe symptom presentation
Change from baseline in Edinburgh Cognitive and Behavioural ALS Screen (ECAS) | 36 weeks for DBPC
  Questionnaire to assesses cognitive and behavioral changes in people with (ALS) through a 136-point test covering language, verbal fluency, executive function, memory, and visuospatial cognitive domains. A lower score indicates worsening of symptoms.
Change from baseline in Edinburgh Cognitive and Behavioural ALS Screen (ECAS) | 36 weeks for OLE
  Questionnaire to assesses cognitive and behavioral changes in people with (ALS) through a 136-point test covering language, verbal fluency, executive function, memory, and visuospatial cognitive domains. A lower score indicates worsening of symptoms.
Change from baseline in ALS Assessment Questionnaire 40 items (ALSAQ-40) | 36 weeks for DBPC
  The ALSAQ40 score is a measure of QoL for patients with ALS. The ALSAQ40 evaluates domains that include physical mobility, activities of daily living (ADL) and independence, eating and drinking, communication, and emotional reactions. A higher score indicates higher disability.
Change from baseline in ALS Assessment Questionnaire 40 items (ALSAQ-40) | 36 weeks for OLE
  The ALSAQ40 score is a measure of QoL for patients with ALS. The ALSAQ40 evaluates domains that include physical mobility, activities of daily living (ADL) and independence, eating and drinking, communication, and emotional reactions. A higher score indicates higher disability.
Change from baseline in Patient Global Impression (PGI) of Improvement | 36 weeks for DBPC
  This will measure all aspects of patient health and improvement or decline. A higher scale indicates greater disability.
Change from baseline in Patient Global Impression (PGI) of Improvement | 36 weeks for OLE
  This will measure all aspects of patient health and improvement or decline. A higher scale indicates greater disability.
Change from baseline in Rasch Overall ALS Disability (ROADS). | 36 weeks for DBPC
  This will measure patient reported outcomes of overall disability. A lower score indicates greater disability.
Change from baseline in Rasch Overall ALS Disability (ROADS). | 36 weeks for OLE
  This will measure patient reported outcomes of overall disability. A lower score indicates greater disability.
Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | 36 weeks for DBPC
  This will assess the safety and tolerability of tazbentetol in of participants with ALS
Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | 36 weeks for OLE
  This will assess the safety and tolerability of tazbentetol in of participants with ALS

OTHER OUTCOMES:
ALSFRS-R total score rate of decline | 36 weeks for DBPC
  To further assess the effect of tazbentetol on the progression of ALS
ALSFRS-R total score rate of decline | 36 weeks for OLE
  To further assess the effect of tazbentetol on the progression of ALS
Proportion of patients alive and survival time | 36 weeks for DBPC
  To further assess the effect of tazbentetol on the progression of ALS
Proportion of patients alive and survival time | 36 weeks for OLE
  To further assess the effect of tazbentetol on the progression of ALS
To compare electroencephalogram (EEG) outcomes of two dose levels of tazbentetol to placebo in participants with ALS | 36 weeks for DBPC
  To measure the change from baseline in EEG delta and power bands at resting state at Weeks 8, 24, and 36

IPD SHARING:
Plan to Share IPD: No